CLINICAL TRIAL: NCT02507089
Title: Tailored Approach to Sleep Health Education: A Community Engaged Approach
Acronym: TASHE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 13-01011; 1R25HL116378-01 (NIH)
Record Dates: First submitted 2015-07-21; First posted 2015-07-23 (Estimated); Last update posted 2019-06-27 (Actual); Status verified 2019-06

CONDITIONS: Healthcare Disparities; Minority Health; Sleep; Sleep Disorders
MeSH Terms: conditions — Sleep Wake Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): In this arm, the participants will receive access to a password protected website that features tailored information and educational materials on sleep health and the signs of sleep disorders such as obstructive sleep apnea (OSA). There will be both text-based information on sleep health and OSA, and also videos depicting narrative stories about patients who have been diagnosed with OSA and sought treatment.
  Interventions: Behavioral: Tailored sleep health education materials.
- Control (Active Comparator): In this arm, participants will receive access to generic sleep educational materials that do not feature linguistic or cultural tailoring to the target population. This arm will include access to the same general information (materials on sleep health, sleep disorder signs and symptoms) but be intended for a general audience.
  Interventions: Behavioral: Generic sleep health education materials.

INTERVENTIONS:
Behavioral: Tailored sleep health education materials. — Tailored sleep health materials.
  Arms: Intervention
Behavioral: Generic sleep health education materials.
  Arms: Control

SUMMARY:
This study aims to develop educational tools and platforms to promote the transfer of sleep health information to blacks to foster adoption of healthful sleep practices.

ELIGIBILITY:
Inclusion Criteria:

* self-reported race/ethnicity as African American, African, Caribbean American or black men and women; ages ≥18 years;
* accessible by telephone; no plans to move away from the region within the year following enrollment;
* consent to participate, which includes permission to release medical record information;
* documented OSA risk based on scores received from the Apnea Risk Evaluation System questionnaire

Exclusion Criteria:

* progressive medical illness in which disability or death is expected within one year;
* impaired cognitive or functional ability which would preclude meaningful participation in the study;
* sleep apnea diagnosis;
* stated intention to move within the same year of enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2014-07; Primary Completion 2017-12 (Actual); Study Completion 2018-02-01 (Actual)

PRIMARY OUTCOMES:
Sleep Hygiene Index | 6 months
Apnea Knowledge/Apnea Belief Scale | 6 months
Self-Efficacy Scale | 6 months
Change Assessment Scale | 6 months

SECONDARY OUTCOMES:
7-Day Physical Activity Recall | 6 months
By-Meal Fruit/Vegetable Intake Screener | 6 months
Rapid Estimate of Adult Literacy in Medicine | 6 months
Medical Outcomes Study Short Form 36 | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Girardin Jean-Louis, PhD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Medical Center, New York, New York, United States

REFERENCES:
- [Derived] Jean-Louis G, Robbins R, Williams NJ, Allegrante JP, Rapoport DM, Cohall A, Ogedegbe G. Tailored Approach to Sleep Health Education (TASHE): a randomized controlled trial of a web-based application. J Clin Sleep Med. 2020 Aug 15;16(8):1331-1341. doi: 10.5664/jcsm.8510. PMID 32329437
- [Derived] Williams NJ, Robbins R, Rapoport D, Allegrante JP, Cohall A, Ogedgebe G, Jean-Louis G. Tailored approach to sleep health education (TASHE): study protocol for a web-based randomized controlled trial. Trials. 2016 Dec 8;17(1):585. doi: 10.1186/s13063-016-1701-x. PMID 27931249